CLINICAL TRIAL: NCT02790242
Title: Registry for Cardiogenic Shock: Utility and Efficacy of Device Therapy
Acronym: RESCUE
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAM2960
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure; Cardiogenic Shock
Keywords: Mechanical Circulatory Support Device (MCSD); ventricular Assist Device (VAD)
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to gather information on patients who have heart failure and are eligible for one of the following two procedures: 1) mechanical support, i.e. ventricular assist device (VAD) or 2) heart transplant. the study seeks to determine which patient populations benefit from heart transplant or ventricular assist device. This will allow to offer the state-of-the-art care to the patients in heart failure.

DETAILED DESCRIPTION:
Cardiogenic shock (CS) develops in the end stage of various etiologies of heart failure and continues to hold high mortality; ranging from 50 to 80%. Expert consensus recommends use of more powerful mechanical circulatory support device (MCSD) in this patient population; however, scientific evidence has been anecdotal relying on mostly single-center small case series and, more fundamentally, because there is no unified definition to grade the severity of the highly heterogeneous condition CS. Well-designed studies are warranted to precisely characterize the various "phenotypes" of CS as well as the role of MCSD in this condition with still excessive mortality.

This multicenter registry will be the first multicenter large-scale registry focused on mechanical circulatory support (MCS) therapy for CS. The fundamental goal of RESCUE is to advance the understanding and application of MCSD in order to improve the persistently dismal survival of patients with CS with the following intents:

1. Elucidate current indication and outcomes of MCSD use in CS.
2. Redefine CS with better description of this disease entity, which will allow better prediction of outcomes, selection of treatment strategy, and comparison and design of studies.
3. Facilitate the refinement of patient selection to maximize outcomes with current and new device options.
4. Improve and expedite new device clinical trials by providing historical control data.
5. Develop consensus "best practice" guidelines to improve clinical management by reducing short and long-term complications of MCSD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who receive any MCSD including Veno-Arterial Extracorporeal Membrane Oxygenation (VA ECMO), surgical VAD, and percutaneous VAD, used to treat CS on or after 9/30/10. Intraaortic balloon pumping (IABP) is not considered an MCSD in this Registry.
* Adult patients who have signed informed consent. For patients who are too ill to give informed consent the health care proxy of the patient or next of kin will be approached for the informed consent.

Exclusion Criteria:

* patients younger than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects include all adult patients who underwent evaluation for MCS for cardiogenic shock. Each adult patient who receives an MCSD at an institution will be screened according to the inclusion and exclusion criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 1089 (Actual)
Dates: Start 2013-11; Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
1-year survival post mechanical circulatory assist device implant | 12 months

SECONDARY OUTCOMES:
survival to discharge post mechanical circulatory assist device implant | until the enrolled patient is discharged. Expected to occur within 90 days of enrollment.
30-day survival post mechanical circulatory assist device implant | 30 days
Number of adverse events during mechanical circulatory assist device support | up to 30-days of weaning from the device.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroo Takayama, MD, PhD, Principal Investigator — Columbia University
Locations (7):
- United States (7):
  - University of Colarodo, Aurora, Colorado
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Newark Beth Israel Medical center, Newark, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hochman JS, Sleeper LA, Webb JG, Sanborn TA, White HD, Talley JD, Buller CE, Jacobs AK, Slater JN, Col J, McKinlay SM, LeJemtel TH. Early revascularization in acute myocardial infarction complicated by cardiogenic shock. SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. N Engl J Med. 1999 Aug 26;341(9):625-34. doi: 10.1056/NEJM199908263410901. PMID 10460813
- [Background] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Fuhrmann J, Bohm M, Ebelt H, Schneider S, Schuler G, Werdan K; IABP-SHOCK II Trial Investigators. Intraaortic balloon support for myocardial infarction with cardiogenic shock. N Engl J Med. 2012 Oct 4;367(14):1287-96. doi: 10.1056/NEJMoa1208410. Epub 2012 Aug 26. PMID 22920912
- [Background] Kirklin JK, Naftel DC, Kormos RL, Stevenson LW, Pagani FD, Miller MA, Baldwin JT, Young JB. Fifth INTERMACS annual report: risk factor analysis from more than 6,000 mechanical circulatory support patients. J Heart Lung Transplant. 2013 Feb;32(2):141-56. doi: 10.1016/j.healun.2012.12.004. PMID 23352390
- [Background] Kirklin JK, Naftel DC, Pagani FD, Kormos RL, Stevenson L, Miller M, Young JB. Long-term mechanical circulatory support (destination therapy): on track to compete with heart transplantation? J Thorac Cardiovasc Surg. 2012 Sep;144(3):584-603; discussion 597-8. doi: 10.1016/j.jtcvs.2012.05.044. Epub 2012 Jul 15. PMID 22795459
- [Background] O'Connor CM, Rogers JG. Evidence for overturning the guidelines in cardiogenic shock. N Engl J Med. 2012 Oct 4;367(14):1349-50. doi: 10.1056/NEJMe1209601. Epub 2012 Aug 26. No abstract available. PMID 22920913